CLINICAL TRIAL: NCT01975675
Title: A Phase 3b, Randomized, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Ledipasvir Fixed-Dose Combination ± Ribavirin in Treatment-Naïve and Treatment-Experienced Japanese Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Efficacy and Safety of Sofosbuvir/Ledipasvir ± Ribavirin in Japanese Participants With Chronic Genotype 1 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0113
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Results first posted 2015-06-26 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2015-06

CONDITIONS: Chronic HCV Infection
MeSH Terms: interventions — Sofosbuvir; ledipasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- LDV/SOF (treatment naive) (Experimental): Treatment-naive participants will receive LDV/SOF for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV (treatment naive) (Experimental): Treatment-naive participants will receive LDV/SOF plus RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF (treatment experienced) (Experimental): Treatment-experienced participants will receive LDV/SOF for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV (treatment experienced) (Experimental): Treatment-experienced participants will receive LDV/SOF plus RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — LDV/SOF 90/400 mg FDC tablet administered orally once daily
  Other Names: GS-7977; PSI-7977; GS-5885
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (≤ 60 kg = 600 mg, > 60 kg to ≤ 80 kg = 800 mg, and ≥ 80 kg = 1000 mg)
  Other Names: Copegus®
  Arms: LDV/SOF+RBV (treatment experienced); LDV/SOF+RBV (treatment naive)

SUMMARY:
This study will evaluate the antiviral efficacy of sofosbuvir (SOF)/ledipasvir (LDV) fixed-dose combination (FDC) tablet with or without ribavirin (RBV) in treatment-naive or treatment-experienced Japanese participants with chronic genotype 1 HCV infection. Participants receive 12 weeks of treatment and continue assessments during a 24-week posttreatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Body weight ≥ 40 kg
* HCV RNA ≥ 10^5 IU/mL at screening

Exclusion Criteria:

* Current or prior history of any clinically-significant illness (other than HCV)
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non-HCV etiology
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Knox, Study Director — Gilead Sciences
Locations (19):
- Japan (19):
  - Ichikawa, Chiba
  - Kurume, Fukuoka
  - Ōgaki, Gifu
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Matsumoto, Nagano
  - Ōmura, Nagasaki
  - Suita, Osaka
  - Izunokuni, Shizuoka
  - Chiyoda-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Musashino, Tokyo
  - Shinjuku, Tokyo
  - Kofu, Yamanashi
  - Akita
  - Chiba
  - Gifu
  - Okayama
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Mizokami M, Yokosuka O, Takehara T, Sakamoto N, Korenaga M, Mochizuki H, Nakane K, Enomoto H, Ikeda F, Yanase M, Toyoda H, Genda T, Umemura T, Yatsuhashi H, Ide T, Toda N, Nirei K, Ueno Y, Nishigaki Y, Betular J, Gao B, Ishizaki A, Omote M, Mo H, Garrison K, Pang PS, Knox SJ, Symonds WT, McHutchison JG, Izumi N, Omata M. Ledipasvir and sofosbuvir fixed-dose combination with and without ribavirin for 12 weeks in treatment-naive and previously treated Japanese patients with genotype 1 hepatitis C: an open-label, randomised, phase 3 trial. Lancet Infect Dis. 2015 Jun;15(6):645-53. doi: 10.1016/S1473-3099(15)70099-X. Epub 2015 Apr 8. PMID 25863559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled study sites in Japan. The first participant was screened on 15 October 2013. The last study visit occurred on 22 August 2014.
Pre-assignment Details: 421 participants were screened.
Groups:
- LDV/SOF (Treatment Naive): Treatment-naive participants received ledipasvir/sofosbuvir (LDV/SOF) 90/400 mg fixed-dose combination (FDC) tablet once daily for up to 12 weeks.
- LDV/SOF+RBV (Treatment Naive): Treatment-naive participants received LDV/SOF 90/400 mg FDC tablet once daily, plus ribavirin (RBV) tablets (600 to 1000 mg daily based on weight) in a divided daily dose for up to 12 weeks.
- LDV/SOF (Treatment Experienced): Treatment-experienced participants received LDV/SOF 90/400 mg FDC tablet once daily for up to 12 weeks.
- LDV/SOF+RBV (Treatment Experienced): Treatment-experienced participants received LDV/SOF 90/400 mg FDC tablet once daily, plus RBV tablets (600 to 1000 mg daily based on weight) in a divided daily dose for up to 12 weeks.
Period: Overall Study
Arm/Group | LDV/SOF (Treatment Naive) | LDV/SOF+RBV (Treatment Naive) | LDV/SOF (Treatment Experienced) | LDV/SOF+RBV (Treatment Experienced)
Started | 83 | 83 | 88 | 87
Completed | 83 | 82 | 88 | 87
Not Completed | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- LDV/SOF (Treatment Naive): Treatment-naive participants received LDV/SOF 90/400 mg FDC tablet once daily for up to 12 weeks.
- LDV/SOF+RBV (Treatment Naive): Treatment-naive participants received LDV/SOF 90/400 mg FDC tablet once daily, plus RBV tablets (600 to 1000 mg daily based on weight) in a divided daily dose for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | LDV/SOF (Treatment Naive) | LDV/SOF+RBV (Treatment Naive) | LDV/SOF (Treatment Experienced) | LDV/SOF+RBV (Treatment Experienced) | Total
Number analyzed (Participants) | 83 | 83 | 88 | 87 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.9) | 59 (10.3) | 61 (8.5) | 59 (8.7) | 59 (9.4)
Age, Customized [Number; unit: participants]
  < 65 years | 60 | 55 | 51 | 63 | 229
  ≥ 65 years | 23 | 28 | 37 | 24 | 112
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 52 | 48 | 199
  Male | 33 | 34 | 36 | 39 | 142
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 83 | 83 | 88 | 87 | 341
Hepatitis C Virus (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.6 (0.48) | 6.6 (0.54) | 6.6 (0.55) | 6.5 (0.54) | 6.6 (0.53)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 6 | 8 | 10 | 13 | 37
  ≥ 800,000 IU/mL | 77 | 75 | 78 | 74 | 304
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 53 | 46 | 33 | 33 | 165
    CT | 29 | 31 | 49 | 51 | 160
    TT | 1 | 6 | 6 | 3 | 16
Cirrhosis Status [Number; unit: participants]
  No | 70 | 71 | 60 | 64 | 265
  Yes | 13 | 12 | 28 | 23 | 76
Response to Prior HCV Treatment [Number; unit: participants]
  Nonresponder | NA — Data not available because treatment-naive participants did not receive prior HCV treatment. | NA — Data not available because treatment-naive participants did not receive prior HCV treatment. | 29 | 28 | NA — Total not calculated because data are not available (NA) in one or more arms.
  Relapse/Breakthrough | NA — Data not available because treatment-naive participants did not receive prior HCV treatment. | NA — Data not available because treatment-naive participants did not receive prior HCV treatment. | 44 | 44 | NA — Total not calculated because data are not available (NA) in one or more arms.
  IFN Intolerant | NA — Data not available because treatment-naive participants did not receive prior HCV treatment. | NA — Data not available because treatment-naive participants did not receive prior HCV treatment. | 15 | 15 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12), Treatment-naive, Noncirrhotic Participants
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Treatment-naive participants in the Full Analysis Set (randomized, received at least 1 dose of study drug, and had chronic genotype 1 (1a, 1b, or mixed 1a/1b) HCV infection) without cirrhosis were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF (Treatment Naive) | LDV/SOF+RBV (Treatment Naive)
Number analyzed (Participants) | 70 | 71
percentage of participants | 100.0 | 97.2
Statistical Analysis 1: Comparison: LDV/SOF (Treatment Naive); Test type: Superiority or Other; p < 0.001, Binomial test — Treatment-naive noncirrhotic participants in the LDV/SOF (treatment naive) group were compared to the adjusted historical SVR null rate of 63% using a two-sided exact one-sample binomial test
Statistical Analysis 2: Comparison: LDV/SOF+RBV (Treatment Naive); Test type: Superiority or Other; p < 0.001, Binomial test — Treatment-naive noncirrhotic participants in the LDV/SOF+RBV (treatment naive) group were compared to the adjusted historical SVR null rate of 63% using a two-sided exact one-sample binomial test

2. Primary Outcome: Percentage of Participants With Sustained Virologic Response at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: as for outcome 1
Time Frame: Posttreatment Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF (Treatment Naive) | LDV/SOF+RBV (Treatment Naive) | LDV/SOF (Treatment Experienced) | LDV/SOF+RBV (Treatment Experienced)
Number analyzed (Participants) | 83 | 83 | 88 | 87
percentage of participants | 100.0 | 96.4 | 100.0 | 100.0
Statistical Analysis 1: Comparison: LDV/SOF (Treatment Naive) vs LDV/SOF+RBV (Treatment Naive); Test type: Superiority or Other; Difference in proportions = -3.6, 95% CI 2-sided [-10.2 to 1.0] — The 95% confidence interval (CI) on the difference in proportions is based on the exact method (standardized statistic and inverting two 1-sided tests)
Statistical Analysis 2: Comparison: LDV/SOF (Treatment Experienced) vs LDV/SOF+RBV (Treatment Experienced); Test type: Superiority or Other; Difference in proportions = 0.0, 95% CI 2-sided [-4.2 to 4.2] — The 95% CI on the difference in proportions is based on the exact method (standardized statistic and inverting two 1-sided tests)

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF (Treatment Naive) | LDV/SOF+RBV (Treatment Naive) | LDV/SOF (Treatment Experienced) | LDV/SOF+RBV (Treatment Experienced)
Number analyzed (Participants) | 83 | 83 | 88 | 87
percentage of participants
  SVR4 | 100.0 | 96.4 | 100.0 | 100.0
  SVR24 | 100.0 | 96.4 | 100.0 | 100.0

4. Secondary Outcome: Percentage of Participants Experiencing Virologic Failure
Description: Virologic failure was defined as
  On-treatment virologic failure:
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  Virologic relapse:
  - Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF (Treatment Naive) | LDV/SOF+RBV (Treatment Naive) | LDV/SOF (Treatment Experienced) | LDV/SOF+RBV (Treatment Experienced)
Number analyzed (Participants) | 83 | 83 | 88 | 87
percentage of participants
  On-treatment virologic failure | 0 | 0 | 0 | 0
  Virologic relapse | 0 | 1.2 | 0 | 0

5. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- LDV/SOF: Participants received LDV/SOF 90/400 mg FDC tablet once daily for up to 12 weeks.
- LDV/SOF+RBV: Participants received LDV/SOF 90/400 mg FDC tablet once daily, plus RBV tablets (600 to 1000 mg daily based on weight) in a divided daily dose for up to 12 weeks.
Arm/Group | LDV/SOF | LDV/SOF+RBV
Number analyzed (Participants) | 171 | 170
percentage of participants | 0 | 1.8

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Arm/Group | LDV/SOF | LDV/SOF+RBV
Serious Adverse Events (participants affected / at risk) | 3/171 | 2/170
Other Adverse Events (participants affected / at risk) | 77/171 | 90/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=171) | LDV/SOF+RBV (N=170)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (N=171) | LDV/SOF+RBV (N=170)
Anaemia (Blood and lymphatic system disorders) | 3 | 23
Nausea (Gastrointestinal disorders) | 5 | 9
Stomatitis (Gastrointestinal disorders) | 6 | 10
Malaise (General disorders) | 9 | 9
Nasopharyngitis (Infections and infestations) | 50 | 40
Headache (Nervous system disorders) | 12 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 13
Rash (Skin and subcutaneous tissue disorders) | 5 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years